CLINICAL TRIAL: NCT03442946
Title: International Nutrition Survey 2018
Acronym: INS2018
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Responsible Party: Principal Investigator, Christian Stoppe, PD Dr. med. Christian Stoppe, University Hospital, Aachen
Other Study IDs: 3CARE_BOÄ_18-001
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cardiovascular Surgery
Keywords: nutrition guidelines; critical care; cardiovascular; nutrition therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- INS: Patients in need of a cardiovascular surgery will be included in this observational study. The focus is on the nutrition therapies provided to these critically ill patients according to institutional or international nutrition guidelines, what ever applies for the participating sites.

SUMMARY:
Malnutrition is common among critically ill patients, and has negative effects on clinical outcomes. Artificial nutrition therapy in the form of enteral or parenteral nutrition is therefore considered an integral part of standard care. While it has long been widely accepted that it is unethical to withhold nutrition therapy from those at risk of malnutrition, we and our collaborators provide first evidence that nutrition practices significantly influence clinically important outcomes such as length of stay, morbidity and mortality in critically ill patients. Among these, cardiac surgery patients are routinely exposed to significant systemic inflammation due to the need for a cardiopulmonary bypass, which triggers a systemic inflammatory response syndrome. As a consequence, the releases of reactive oxygen and nitrogen species as well as pro-inflammatory cytokines lead to life-threatening complications in cardiac surgical patients. For such patients, aggressive life-sustaining therapies are needed while their organs recover.

Besides, underfeeding is a major issue in this specific patient population. Often nutrition starts late and reaches only low nutrition adequacy. Recent data from our collaborators suggest that providing at least 80% of prescribed amounts of protein and energy is associated with improved clinical outcomes. Achieving this threshold of 80% of prescribed amounts of protein has been shown to be associated with reduced mortality in "at-risk" ICU patients and is more important than achieving energy goals. Despite these benefits, enteral or parenteral feeding should always be adopted with caution, as nutrition practices themselves are not per se without adverse effects or risks. Making decisions regarding the most effective and safe means of feeding patients in the ICU can be challenging, and consequently considerable variation exists in nutrition practices in this setting, whereas no guidelines yet exists specific of cardiac surgery patients.

Clinical Practice Guidelines (CPGs) are "systematically developed statements to assist practitioner and patient decisions about appropriate health care for specific clinical circumstances", and therefore aid in the implementation of evidence-based medicine. The Canadian Clinical Practice Guidelines for Nutrition Therapy in Mechanically Ventilated, Critically Ill Adult Patients published in 2003 by our close collaborator Prof Heyland and most recently updated in 2015, sought to improve nutrition practices in ICUs across Canada and worldwide by providing guidance to select and deliver the most appropriate form of nutrition therapy at the appropriate time via the most appropriate route. A validation study prior to the widespread dissemination of the Canadian Critical Care Nutrition CPGs concluded that adoption of the recommendations should lead to improved nutrition practices and potentially to better patient outcomes [24]. To change clinical practice, attention must extend beyond initial development to guideline implementation, dissemination and evaluation. Implementation strategies will vary by ICU, health care system and region and should be guided by local factors including the ICU's barriers and facilitators to following best practice. Evaluating and monitoring nutrition performance and focussing on different groups of critically ill patients, should be part of an on-going improvement strategy to improve nutrition care and clinical outcome. The few studies regarding the process of knowledge translation conducted in the ICU setting have demonstrated by our collaborators that guidelines and guideline implementation strategies improve the processes, outcomes, and the costs of caring for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients undergoing cardiac surgery
* Mechanically ventilated within 48 hours of ICU admission
* Stay on ICU > 72 hours

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in need of a cardiovascular surgery and meeting the inclusion criteria are considered to be eligible for this study.
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in nutrition adequacy in the ICU | day 1, day 2, day 3, day 4, day 5, day 6, day 7, day 8, day 9, day 10, day 11, day 12
  Adequacy of nutrition (an indicator of overall performance) will be calculated as the amount of calories or protein received (from either enteral (EN) or appropriate parenteral nutrition (PN) but not oral) plus propofol, divided by the amount prescribed as per the baseline assessment and expressed as a percentage. Days without EN or PN will be included and counted as 0% adequacy. Days after permanent progression to exclusive oral intake will be excluded from the calculation of nutritional adequacy. We arbitrarily selected >80% nutritional adequacy as an indicator of high performance.

CONTACTS AND LOCATIONS:
Locations (5):
- University of Utah Medical Center, Salt Lake City, Utah, United States
- Sunnybrook Health Sciences Centre, Toronto, Canada
- University hospital RWTH Aachen, Aachen, Germany
- Rajaie Cardiovascular, Medical and Research Center, Tehran, Iran
- Meshalkin National Medical Research Center, Novosibirsk, Russia

REFERENCES:
- [Result] Giner M, Laviano A, Meguid MM, Gleason JR. In 1995 a correlation between malnutrition and poor outcome in critically ill patients still exists. Nutrition. 1996 Jan;12(1):23-9. doi: 10.1016/0899-9007(95)00015-1. PMID 8838832
- [Result] Heyland DK. Nutritional support in the critically ill patients. A critical review of the evidence. Crit Care Clin. 1998 Jul;14(3):423-40. doi: 10.1016/s0749-0704(05)70009-9. PMID 9700440
- [Result] Heyland DK, Novak F, Drover JW, Jain M, Su X, Suchner U. Should immunonutrition become routine in critically ill patients? A systematic review of the evidence. JAMA. 2001 Aug 22-29;286(8):944-53. doi: 10.1001/jama.286.8.944. PMID 11509059
- [Result] Heyland DK, Drover JW, Dhaliwal R, Greenwood J. Optimizing the benefits and minimizing the risks of enteral nutrition in the critically ill: role of small bowel feeding. JPEN J Parenter Enteral Nutr. 2002 Nov-Dec;26(6 Suppl):S51-5; discussion S56-7. doi: 10.1177/014860710202600608. PMID 12405623
- [Result] Novak F, Heyland DK, Avenell A, Drover JW, Su X. Glutamine supplementation in serious illness: a systematic review of the evidence. Crit Care Med. 2002 Sep;30(9):2022-9. doi: 10.1097/00003246-200209000-00011. PMID 12352035
- [Result] Gramlich L, Kichian K, Pinilla J, Rodych NJ, Dhaliwal R, Heyland DK. Does enteral nutrition compared to parenteral nutrition result in better outcomes in critically ill adult patients? A systematic review of the literature. Nutrition. 2004 Oct;20(10):843-8. doi: 10.1016/j.nut.2004.06.003. PMID 15474870
- [Result] Stoppe C, Meybohm P, Coburn M, Goetzenich A. [Cardioprotection in cardiac surgical patients : Everything good comes from the heart]. Anaesthesist. 2016 Mar;65(3):169-82. doi: 10.1007/s00101-016-0141-z. German. PMID 26915019
- [Result] Kim BS, Jacobs D, Emontzpohl C, Goetzenich A, Soppert J, Jarchow M, Schindler L, Averdunk L, Kraemer S, Marx G, Bernhagen J, Pallua N, Schlemmer HP, Simons D, Stoppe C. Myocardial Ischemia Induces SDF-1alpha Release in Cardiac Surgery Patients. J Cardiovasc Transl Res. 2016 Jun;9(3):230-238. doi: 10.1007/s12265-016-9689-x. Epub 2016 Apr 7. PMID 27055858
- [Result] Dreymueller D, Goetzenich A, Emontzpohl C, Soppert J, Ludwig A, Stoppe C. The perioperative time course and clinical significance of the chemokine CXCL16 in patients undergoing cardiac surgery. J Cell Mol Med. 2016 Jan;20(1):104-15. doi: 10.1111/jcmm.12708. Epub 2015 Oct 23. PMID 26499307
- [Result] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Result] Drover JW, Cahill NE, Kutsogiannis J, Pagliarello G, Wischmeyer P, Wang M, Day AG, Heyland DK. Nutrition therapy for the critically ill surgical patient: we need to do better! JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):644-52. doi: 10.1177/0148607110372391. PMID 21097764
- [Result] Rahman A, Hasan RM, Agarwala R, Martin C, Day AG, Heyland DK. Identifying critically-ill patients who will benefit most from nutritional therapy: Further validation of the "modified NUTRIC" nutritional risk assessment tool. Clin Nutr. 2016 Feb;35(1):158-162. doi: 10.1016/j.clnu.2015.01.015. Epub 2015 Jan 28. PMID 25698099
- [Result] Heyland DK, Cahill N, Day AG. Optimal amount of calories for critically ill patients: depends on how you slice the cake! Crit Care Med. 2011 Dec;39(12):2619-26. doi: 10.1097/CCM.0b013e318226641d. PMID 21705881
- [Result] Nicolo M, Heyland DK, Chittams J, Sammarco T, Compher C. Clinical Outcomes Related to Protein Delivery in a Critically Ill Population: A Multicenter, Multinational Observation Study. JPEN J Parenter Enteral Nutr. 2016 Jan;40(1):45-51. doi: 10.1177/0148607115583675. Epub 2015 Apr 21. PMID 25900319
- [Result] Mentec H, Dupont H, Bocchetti M, Cani P, Ponche F, Bleichner G. Upper digestive intolerance during enteral nutrition in critically ill patients: frequency, risk factors, and complications. Crit Care Med. 2001 Oct;29(10):1955-61. doi: 10.1097/00003246-200110000-00018. PMID 11588461
- [Result] Heyland DK, MacDonald S, Keefe L, Drover JW. Total parenteral nutrition in the critically ill patient: a meta-analysis. JAMA. 1998 Dec 16;280(23):2013-9. doi: 10.1001/jama.280.23.2013. PMID 9863853
- [Result] Heyland DK, Schroter-Noppe D, Drover JW, Jain M, Keefe L, Dhaliwal R, Day A. Nutrition support in the critical care setting: current practice in canadian ICUs--opportunities for improvement? JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):74-83. doi: 10.1177/014860710302700174. PMID 12549603
- [Result] Mead P. Clinical guidelines: promoting clinical effectiveness or a professional minefield? J Adv Nurs. 2000 Jan;31(1):110-6. doi: 10.1046/j.1365-2648.2000.01254.x. PMID 10632799
- [Result] Miller M, Kearney N. Guidelines for clinical practice: development, dissemination and implementation. Int J Nurs Stud. 2004 Sep;41(7):813-21. doi: 10.1016/j.ijnurstu.2003.09.005. PMID 15288803
- [Result] Heyland DK, Dhaliwal R, Drover JW, Gramlich L, Dodek P; Canadian Critical Care Clinical Practice Guidelines Committee. Canadian clinical practice guidelines for nutrition support in mechanically ventilated, critically ill adult patients. JPEN J Parenter Enteral Nutr. 2003 Sep-Oct;27(5):355-73. doi: 10.1177/0148607103027005355. PMID 12971736
- [Result] Heyland DK, Dhaliwal R, Day A, Jain M, Drover J. Validation of the Canadian clinical practice guidelines for nutrition support in mechanically ventilated, critically ill adult patients: results of a prospective observational study. Crit Care Med. 2004 Nov;32(11):2260-6. doi: 10.1097/01.ccm.0000145581.54571.32. PMID 15640639
- [Result] Pilon CS, Leathley M, London R, McLean S, Phang PT, Priestley R, Rosenberg FM, Singer J, Anis AH, Dodek PM. Practice guideline for arterial blood gas measurement in the intensive care unit decreases numbers and increases appropriateness of tests. Crit Care Med. 1997 Aug;25(8):1308-13. doi: 10.1097/00003246-199708000-00016. PMID 9267942
- [Result] Pitimana-aree S, Forrest D, Brown G, Anis A, Wang XH, Dodek P. Implementation of a clinical practice guideline for stress ulcer prophylaxis increases appropriateness and decreases cost of care. Intensive Care Med. 1998 Mar;24(3):217-23. doi: 10.1007/s001340050553. PMID 9565802
- [Result] Sinuff T, Cook DJ, Randall J, Allen CJ. Evaluation of a practice guideline for noninvasive positive-pressure ventilation for acute respiratory failure. Chest. 2003 Jun;123(6):2062-73. doi: 10.1378/chest.123.6.2062. PMID 12796190
- [Result] Martin CM, Doig GS, Heyland DK, Morrison T, Sibbald WJ; Southwestern Ontario Critical Care Research Network. Multicentre, cluster-randomized clinical trial of algorithms for critical-care enteral and parenteral therapy (ACCEPT). CMAJ. 2004 Jan 20;170(2):197-204. PMID 14734433
- [Result] Burns SM, Earven S, Fisher C, Lewis R, Merrell P, Schubart JR, Truwit JD, Bleck TP; University of Virginia Long Term Mechanical Ventilation Team. Implementation of an institutional program to improve clinical and financial outcomes of mechanically ventilated patients: one-year outcomes and lessons learned. Crit Care Med. 2003 Dec;31(12):2752-63. doi: 10.1097/01.CCM.0000094217.07170.75. PMID 14668611
- [Result] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094
- [Result] Compher C, Chittams J, Sammarco T, Nicolo M, Heyland DK. Greater Protein and Energy Intake May Be Associated With Improved Mortality in Higher Risk Critically Ill Patients: A Multicenter, Multinational Observational Study. Crit Care Med. 2017 Feb;45(2):156-163. doi: 10.1097/CCM.0000000000002083. PMID 28098623
- [Result] Heyland DK, Dhaliwal R, Wang M, Day AG. The prevalence of iatrogenic underfeeding in the nutritionally 'at-risk' critically ill patient: Results of an international, multicenter, prospective study. Clin Nutr. 2015 Aug;34(4):659-66. doi: 10.1016/j.clnu.2014.07.008. Epub 2014 Jul 19. PMID 25086472
- [Result] Heyland DK, Heyland RD, Cahill NE, Dhaliwal R, Day AG, Jiang X, Morrison S, Davies AR. Creating a culture of clinical excellence in critical care nutrition: the 2008 "Best of the Best" award. JPEN J Parenter Enteral Nutr. 2010 Nov-Dec;34(6):707-15. doi: 10.1177/0148607110361901. PMID 21097771